CLINICAL TRIAL: NCT00755404
Title: Phase 2 Study of the Effect of a Peritoneal Dialysis Solution Containing Glucose (1.5%) and L-Carnitine (0.1%) on Insulin Sensitivity in Patients on Continuous Ambulatory Peritoneal Dialysis
Brief Title: Effect of an L-Carnitine-Containing Peritoneal Dialysis (PD) Solution on Insulin Sensitivity in Diabetic Patients on Continuous Ambulatory Peritoneal Dialysis (CAPD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-003-05
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2013-03

CONDITIONS: End Stage Renal Disease; Diabetes
Keywords: Peritoneal dialysis; L-carnitine; Diabetes; Glucose homeostasis; Dyslipidemia
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: PD Solution
- B (Experimental)
  Interventions: Drug: PD solution containing L-carnitine

INTERVENTIONS:
Drug: PD Solution — Instillation of PD solutions containing Glucose (1.5 or 2.5%, w/v) for the diurnal exchanges, and 1 PD solution containing icodextrin (7.5 w/v) for nocturnal exchange. PD solutions are instilled for 180 days.
  Arms: A
Drug: PD solution containing L-carnitine — Instillation of PD solutions containing Glucose (1.5 or 2.5%, w/v) and L-carnitine (0.1%, w/v) for the diurnal exchanges, and 1 PD solution containing icodextrin (7.5 w/v) for nocturnal exchanges. PD solutions are instilled for 180 days.
  Arms: B

SUMMARY:
The current study is initiated in order to assess the impact of a PD solution containing L-carnitine on insulin sensitivity evaluated by measuring insulin requirement.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Have a diagnosis of ESRD and have been on Continuous Ambulatory Peritoneal Dialysis (CAPD) for at least 3 months
3. Have Type 2 Diabetes, diagnosed according to American Diabetes Association (fasting glucose ≥126 mg/dl and 2 h glucose at OGTT ≥200 mg/dl), and treated with multiple daily insulin injection or with HbA1c > 8.5% (No oral antidiabetic)
4. Be in a stable clinical condition during the four weeks immediately prior to Screening Period as demonstrated by medical history, physical examination and laboratory testing
5. Have a blood hemoglobin concentration above 8,5 g/100ml (data will be verified with Investigators)
6. Have not experienced peritonitis episodes in the last 3 months
7. Be treated with Extraneal (nocturnal exchange bag solution) for at least 1 month
8. Be treated with 3 diurnal exchange bag solutions (solution bags with 1.5% or 2.5% glucose) and one nocturnal exchange bag solution (Extraneal)
9. Have Kt/V urea measurement > 1.7 per week in a previous test performed within 3 months that should be confirmed at Baseline Visit
10. Have a minimum weekly creatinine clearance of 45 litres in a previous test performed within 6 months that should be confirmed at Baseline Visit
11. Have a D/P Creatinine ratio at Peritoneal Equilibration Test (PET) between 0.50 and 0.81 in a previous test performed within 6 months that should be confirmed at Baseline Visit
12. Have a D/P Glucose ratio at Peritoneal Equilibration Test (PET) between 0.26 and 0.49 in a previous test performed within 6 months that should be confirmed at Baseline Visit
13. Be treated by the participating clinical Investigator for a period of at least three months
14. Have understood and signed the Informed Consent Form.

Exclusion Criteria:

1. Have a history of drug or alcohol abuse in the six months prior to entering the protocol
2. Type 2 Diabetic patients under oral antidiabetic treatment with HbA1C < 8.5%
3. Be in treatment with androgens
4. Have clinically significant abnormal liver function test (SGOT, SGPT, and gamma-GT > 2 times the upper normal limit)
5. Have acute infectious conditions (i.e.: pulmonary infection, acute hepatitis, high or low urinary tract infections, renal parenchymal infection, pericarditis, etc)
6. Have a history of congestive heart failure and clinically significant arrhythmia
7. Have an history of epilepsy or any CNS disease
8. Have malignancy within the past 5 years, including lymphoproliferative disorders
9. Have any medical condition that, in the judgment of the Investigator, would jeopardize the patient's safety following exposure to study drug
10. Have a history of L-Carnitine therapy or use in the month prior to entering the protocol
11. Have used any investigational drug in the 3 months prior to entering the protocol
12. Be in pregnancy, lactation, fertility age without protection against pregnancy by adequate contraceptive means

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of L-Carnitine containing PD solution on insulin sensitivity evaluated by measuring insulin requirement | time 0, 6 months

SECONDARY OUTCOMES:
To assess the efficacy of L-Carnitine containing PD solution on plasma lipids and lipoprotein profile | 4 weeks, time 0, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
To assess the efficacy of L-Carnitine containing PD solution on hematological parameters (hemoglobin and EPO requirements) | 2 weeks, time 0, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco P Schena, MD, Principal Investigator — University of Bari; Arduino Arduini, MD, Study Director — Iperboreal Pharma Srl
Locations (8):
- Italy (8):
  - Renal, Dialysis and Transplant Unit, University of Bari, Bari
  - Division of Nephrology, University of "G. d'Annunzio", Chieti
  - Nephrology and Dialysis Unit, Desio Hospital, Desio
  - Nephrology and Dialysis Unit, "Maria SS dello Splendore" Hospital, Giulianova
  - Division of Nephrology and Dialysis, Ospedale Policlinico Maggiore, Milan
  - Nephrology and Dialysis Unit, "G. Bernabeo" Hospital, Ortona
  - Renal Unit, Policlinico MultiMedica, Sesto San Giovanni
  - Division of Nephrology and Dialysis, "Mazzini" Hospital, Teramo